CLINICAL TRIAL: NCT00006448
Title: Spinal Cord Injury (SCI) and Amputation Pain Prevention and Treatment
Brief Title: Treatment of Chronic Pain After Spinal Cord Injury (SCI) or Amputation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NICHD-0108; 5P01HD033989-05 (NIH)
Record Dates: First submitted 2000-11-04; First posted 2000-11-06 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2003-03

CONDITIONS: Spinal Cord Injuries; Amputation, Traumatic; Pain
Keywords: Spinal cord injury; Amputation; Pain management
MeSH Terms: conditions — Spinal Cord Injuries; Amputation, Traumatic; Pain; Agnosia | interventions — Cognitive Behavioral Therapy; Physical Therapy Modalities; Methadone

INTERVENTIONS:
Behavioral: cognitive therapy
Procedure: Physical Therapy
Drug: Methadone

SUMMARY:
Pain is a major problem for people after spinal cord injuries and amputations. This is a study to test how pain is affected by adding methadone to a six-week program of weekly physical therapy, relaxation training and counseling. Individuals who qualify for this study will receive a comprehensive medical and physical therapy evaluation.

DETAILED DESCRIPTION:
Pain has a major impact on the functioning of individuals with spinal cord injuries and individuals with amputations. This double-masked randomized trial to evaluate the utility of a combination of psychological intervention and physical therapy in order to improve pain reduction, increase physical functioning and quality of life for patients with pain associated with spinal cord injuries or amputations will compare the effect of a 6 week program of physical therapy and cognitive-behavioral therapy with methadone to one without methadone (n = 400). Secondary outcomes are to evaluate the maintenance of effects of the combined intervention and to evaluate the usefulness of a course of opioid therapy compared to active placebo medication. Based on the sample size, all measures have greater than 0.7 power to detect major within group differences at posttreatment, 6-month follow-up, and 12-month follow-up (taking into account a 15% attrition rate, alpha .05). Patients who qualify for this study will receive a comprehensive medical and physical therapy evaluation at baseline. Outcome will be assessed by the physician, psychiatrist and physical therapist who are all masked both to the treatment condition and therapy. Pain is assessed through self-report (measures include pain inventories) and clinical interview.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with spinal cord injury or amputation, who have persistent pain of three months or longer duration.

Exclusion Criteria:

* Pregnant women
* Allergy to latex, methadone, or diphenhydramine
* Surgery planned
* History of substance abuse in past two years
* History of major psychiatric disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 1996-08; Primary Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Rudy, Ph.D., Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburg Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- See also: Click here for more information about the National Institute of Child Health and Human Development (NICHD). — http://www.nichd.nih.gov